CLINICAL TRIAL: NCT02115165
Title: A Prospective Phase II Trial of Cabazitaxel in Male Patients With Chemotherapy Pre-treated Metastatic Nonseminomatous Germ-cell Tumors
Brief Title: A Prospective Study of Cabazitaxel in Patients With Non Seminomatous Germ-cell Tumors
Acronym: CABA-GCT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-000286-36; 2012/1950 (Other: CSET number)
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Non-seminomatous Germ-cell Tumors
MeSH Terms: conditions — Nonseminomatous germ cell tumor | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental)
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — On Day 1 of each cycle, patients will receive cabazitaxel at a dose of 25 mg/m², administered by IV route in 1 hour

SUMMARY:
Cabazitaxel is a new generation taxane with a high capacity for blood-brain barrier crossing and limited peripheral neuro-toxicity, two major potential advantages in patients with advanced NSGCTs.

Cabazitaxel has a broader in vitro spectrum of activity than docetaxel. Taxanes have demonstrated activity in pre-treated GCTs and are now part of standard treatment, but cabazitaxel has not yet been tested in patients with NSGCT.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 15 years or older
* Evidence of advanced NSGCT documented either by pathology or by elevated tumor markers (AFP or hCG) and a compatible clinical presentation
* Primary site located in either the testis, the retroperitoneum or the mediastinum
* Progressive disease after at least 2 lines of chemotherapy for advanced NSGCT (ie, non-stage I)
* In case of brain metastases, confirm that patients should be stable / controlled with corticosteroid/anti seizures agents
* No other progressive carcinoma within previous the 5 years, except for basal-cell carcinoma of the skin
* Life expectancy >/= 3 months
* Adequate hematologic function :
* Hemoglobin >/= 10.0 g/dL
* Absolute neutrophil count >/= 1.5 x 10 ^ 9/L,
* Platelet count >/= 100 x 10 ^ 9/L,
* Adequate organ function
* Serum creatinine < 1.5 x ULN. If serum creatinine 1.0 - 1.5 x ULN, creatinine clearance calculated (or measured) according to CKD-EPI formula (see Appendix B) > 60 mL/min
* AST/SGOT and ALT/SGPT </= 1.5 x ULN
* Bilirubin </= 1.5 x ULN
* Information delivered to patient and informed consent form signed by the patient or his legal representative
* Patient affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

* Patients receiving anti cancer therapy within 4 weeks prior to enrolment
* Previous radiotherapy within 4 weeks prior to enrolment
* Serious uncontrolled concurrent medical illness
* History of severe hypersensitivity reaction (>/= grade 3) to polysorbate 80 containing drugs or to other taxanes
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P450 3A4/5 (see Appendix A). A one week wash-out period is necessary for patients who are already on these treatments.
* Patient with reproductive potential not implementing accepted and effective method of contraception for up to 6 months after the last dose of cabazitaxel.
* Active Grade >/= 3 peripheral neuropathy
* Patients who have had a major surgery within 4 last weeks prior enrolment
* Uncontrolled cardiac arrhythmias, angina pectoris, and/or hypertension. History of congestive heart failure (NYHA III or IV) or myocardial infarction within last 6 months is also not allowed

Min Age: 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Favorable response | Assessed every 6 weeks from start of treatment up to 72 months
  To evaluate the favorable response rate of cabazitaxel treatment in patients with highly-pretreated nonseminomatous germ-cell tumors (NSGCT)

SECONDARY OUTCOMES:
Response rate on brain metastases | Assessed every 6 weeks after treatment start up to 72 months
  MRI of the brain every 6 weeks only in case of brain metastases detected at baseline and for all patients at the end of the study.
  Evaluation will be made using RECIST V1.1
Progression free survival | Assessed every 6 weeks from treatment start to progression up to 72 months
Overall survival | Assessed every 3 weeks after treatment start up to 72 months

CONTACTS AND LOCATIONS:
Overall Officials: Karim FIZAZI, MD-PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val de Marne, France